CLINICAL TRIAL: NCT04937478
Title: Correlation of Ultrafiltered Volume (UFV) During Hemodialysis With a New Battery Powered, Body Worn Electronic Patch Measuring Bioimpedance.
Brief Title: Correlation of Ultrafiltered Volume (UFV) to Bioimpedance Changes
Acronym: CTR006
Status: Completed | Type: Observational
Sponsor: Mode Sensors AS (Industry)
Collaborators: St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: CTR006 DELAGE 2
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hemodialysis, Ultrafiltration, Bioimpedance
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum:
  * osmolality
  * hemoglobin
  * platelets
  * sodium
  * potassium
  * creatinine
  * urea
  * glucose
  * magnesium
  * albumin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis patients: Patients who undergo hemodialysis in hospital every two to three days.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Only observational study, no intervention.

SUMMARY:
Patient submitted to hemodialysis are followed through a dialysis - interim - dialysis cycle.

No intervention is done. Additional blood tests and clinical tests are used as pseudo-endpoints. Correlation is made to ultrafiltrated volume (UFV).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for hemodialysis
* signed Informed Consent Form

Exclusion Criteria:

* acute intercurrent disease,
* subjects with known hypersensitivity to plasters (adhesive or gel).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with hemodialysis for survival.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation between ultrafiltered volume (UFV) and measured bioimpedance change | During hemodialysis
  A change in measured thoracic bioimpedance is expected to correlate to UFV

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Levanger Hospital, Levanger
  - St Olavs university hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared